CLINICAL TRIAL: NCT05174312
Title: Fluid Management of Acute Decompensated Heart Failure Subjects Treated With Reprieve Decongestion Management System (DMS) - FASTR Trial
Brief Title: Fluid Management of Acute Decompensated Heart Failure Subjects Treated With Reprieve Decongestion Management System (DMS)
Acronym: FASTR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reprieve Cardiovascular, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCV-0006
Record Dates: First submitted 2021-12-06; First posted 2021-12-30 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Acute Decompensated Heart Failure
MeSH Terms: interventions — Diuretics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Reprieve Decongestion Management System (Experimental): Subjects randomized to Reprieve System will receive personalized and optimized diuretic and saline infusion using the study device during the course of the treatment.
  Interventions: Device: Reprieve Decongestion Management System
- Optimal Diuretic Therapy (Active Comparator): Sites will consider best practices of optimal diuretic dosing such as those demonstrated in recent randomized trials (DOSE, ADVOR, CLOROTIC) for patients randomized to control arm of the trial.
  Interventions: Drug: Diuretic

INTERVENTIONS:
Device: Reprieve Decongestion Management System — The Reprieve Decongestion Management System, or Reprieve DMS, is a hospital bedside fluid management console designed to provide personalized and automated infusion of the IV diuretic furosemide and physiological saline in response to the patient's real-time urine output to safely and rapidly decongest patients suffering from Acute Decompensated Heart Failure.
  Arms: Reprieve Decongestion Management System
Drug: Diuretic — Best practices of optimal diuretic dosing such as those demonstrated in recent randomized trials (DOSE, ADVOR, CLOROTIC).
  Arms: Optimal Diuretic Therapy

SUMMARY:
The objective of this study is to prospectively compare decongestive therapy administered by the Reprieve DMS system to Optimal Diuretic Therapy (ODT) in the treatment of patients diagnosed with acute decompensated heart failure (ADHF). The main objective is to determine if the Reprieve DMS can more efficiently decongest ADHF patients in comparison to Control Therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized with a diagnosis of heart failure as defined by the presence of at least 1 symptom AND 1 sign.
2. ≥10 pounds (4.5 kg) above dry weight either by historical weights or as estimated by health care provider.
3. Prior use of loop diuretics within 30 says prior to admission.
4. ≥ 18 years of age able to provide informed consent and comply with study procedures.

Exclusion Criteria:

1. Inability to place Foley catheter or IV catheter.
2. Hemodynamic instability.
3. Dyspnea due primarily to non-cardiac causes.
4. Acute infection with evidence of systemic involvement.
5. Estimated glomerular filtration rate (eGFR) < 20 ml/min/1.73m2 calculated using the MDRD equation or current use of renal replacement therapy.
6. Significant left ventricular outflow obstruction, uncorrected complex congenital heart disease, severe stenotic valvular disease, infiltrative or constrictive cardiomyopathy, acute myocarditis, type 1 acute myocardial infarction requiring treatment, or any other pathology that, in the opinion of the investigator, would make aggressive diuresis poorly tolerated.
7. Inability to follow instructions or comply with follow-up procedures.
8. Other concomitant disease or condition that investigator deems unsuitable for the study, including drug or alcohol abuse or psychiatric, behavioral or cognitive disorders, sufficient to interfere with the patient's ability to understand and comply with the study instructions or follow-up procedures.
9. Severe electrolyte abnormalities.
10. Presence of active coronavirus disease 2019 (COVID-19) infection.
11. Enrollment in another interventional trial during the index hospitalization.
12. Inability to return for follow-up study visits.
13. Life expectancy less than 3 months.
14. Women who are pregnant or intend to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Total urine sodium output | 24 hours post-treatment initiation
  Primary efficacy endpoint is total urine sodium output at 24 hours post-treatment initiation.
Clinically significant acute kidney injury, severe electrolyte abnormality, symptomatic hypotension or hypertensive emergency. | Through study completion, an average of 90 days
  Primary safety endpoint includes clinically significant acute kidney injury defined as KDIGO stage 2 or greater AKI [≥ doubling of baseline serum creatinine or use of renal replacement therapy (RRT)], severe electrolyte abnormality (serum potassium <3.0 mEq/L, magnesium <1.3 mEq/L or sodium <125 mEq), symptomatic hypotension or hypertensive emergency.

SECONDARY OUTCOMES:
Net fluid loss | End of treatment, an average of 72 hours
  Difference in the amount of net fluid removed during primary treatment
Time on loop diuretics | End of treatment, an average of 72 hours
  Total time on loop diuretics during primary treatment

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Eastern Shore Research Institute, Fairhope, Alabama
  - University of California Irvine, Irvine, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Trinity Health Ann Arbor Hospital, Ypsilanti, Michigan
  - St. Louis VA, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Duke University Hospital, Durham, North Carolina
  - Cone Health, Greensboro, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - The Lindner Research Center at Christ Hospital, Cincinnati, Ohio
  - Ohio State University Hospital, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health, Columbia, South Carolina
  - Ascension Texas Cardiovascular, Austin, Texas
  - Baylor Scott & White, Dallas, Texas
  - University of Vermont Medical Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No